CLINICAL TRIAL: NCT04339595
Title: A Phase IV Interventional Study to Assess the Disease-Modifying Effect of Long-Term Treatment With Tildrakizumab in Adult Patients With Moderate-To-Severe Plaque Psoriasis (MODIFY)
Brief Title: Long-Term Treatment Effect With Tildrakizumab in Participants With Plaque Psoriasis
Acronym: MODIFY
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low Recruitment
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-14745-44; 2019-003218-15 (EudraCT Number)
Record Dates: First submitted 2020-03-25; First posted 2020-04-09 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Plaque Psoriasis
Keywords: Human Antibody; Interleukin (IL) -23p19; Tildrakizumab; Moderate-To-Severe Plaque Psoriasis
MeSH Terms: interventions — tildrakizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tildrakizumab (Experimental)
  Interventions: Biological: Tildrakizumab

INTERVENTIONS:
Biological: Tildrakizumab — Participants who have participated and completed the long-term extension phase of the reSURFACE 2 study (NCT01729754) and 12 weeks after the last Tildrakizumab dose will be included in the present study. Participants will not receive any study medication during the present study. Participants will remain in the study for 96 weeks or until they initiate any systemic therapy for psoriasis (including phototherapy), whichever occurs first.

SUMMARY:
The purpose of this study is to evaluate the psoriasis disease control over time in participants who had received Tildrakizumab for at least the last 5 years and have discontinued it and to describe blood and skin inflammatory biomarkers and its correlation disease relapse.

ELIGIBILITY:
Inclusion Criteria:

* Participants provide signed written informed consent prior to perform any study-related activity
* Participants has completed the long-term extension of the reSURFACE 2 study

Exclusion Criteria:

* Participants unable to comply with the requirements of the study
* Participants who in the opinion of the investigator should not participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Presence of Blood Inflammatory Biomarkers at Baseline | Baseline
  Inflammatory biomarkers will be assessed using blood serum/plasma sample collected for local safety analysis.
Number of Participants with Presence of Blood Inflammatory Biomarkers at Week 12 | Week 12
  Inflammatory biomarkers will be assessed using blood serum/plasma sample collected for local safety analysis.
Number of Participants with Presence of Blood Inflammatory Biomarkers at Week 24 | Week 24
  Inflammatory biomarkers will be assessed using blood serum/plasma sample collected for local safety analysis.
Number of Participants with Presence of Blood Inflammatory Biomarkers at Week 36 | Week 36
  Inflammatory biomarkers will be assessed using blood serum/plasma sample collected for local safety analysis.
Number of Participants with Presence of Blood Inflammatory Biomarkers at Week 48 | Week 48
  Inflammatory biomarkers will be assessed using blood serum/plasma sample collected for local safety analysis.
Number of Participants with Presence of Blood Inflammatory Biomarkers at Week 60 | Week 60
  Inflammatory biomarkers will be assessed using blood serum/plasma sample collected for local safety analysis.
Number of Participants with Presence of Blood Inflammatory Biomarkers at Week 72 | Week 72
  Inflammatory biomarkers will be assessed using blood serum/plasma sample collected for local safety analysis.
Number of Participants with Presence of Blood Inflammatory Biomarkers at Week 84 | Week 84
  Inflammatory biomarkers will be assessed using blood serum/plasma sample collected for local safety analysis.
Number of Participants with Presence of Blood Inflammatory Biomarkers at Week 96/End of Study (EOS) | Week 96/End of study (EOS)
  Inflammatory biomarkers will be assessed using blood serum/plasma sample collected for local safety analysis.
Number of Participants with Presence of Skin Inflammatory Biomarkers at Baseline | Baseline
  Inflammatory biomarkers will be assessed using a small piece of 4 millimeter (mm) of skin biopsy sample collected at Baseline (stored in RNAlater solution).
Number of Participants with Presence of Skin Inflammatory Biomarkers at Week 48 or End of Study (EOS) | up to Week 48
  Inflammatory biomarkers will be assessed using a small piece of 4 millimeter (mm) of skin biopsy sample collected at Week 48 or until the date of initiation of any systemic therapy including phototherapy whichever comes first (EOS) (stored in RNAlater solution).
Percentage of Participants Who Experienced Psoriasis Relapse | Baseline up to Week 96/ End of study (EOS)
  Psoriasis Area and Severity Index (PASI) is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and scaling on a scale range from 0 (no symptoms) to 4 (very marked), together with the percentage (%) of the area affected, rated on a scale from 0 (0%) to 6 (90-100%). PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 (no psoriasis) to 72 (the most severe disease). Relapse is defined using the following thresholds: PASI greater than (>) 3 (participants who had a PASI lesser than or equal to [<=] 3 at baseline); PASI > 5 (participants who had a PASI <= 5 at baseline); DLQI > 5 (participants who had a DLQI <= 5 at baseline); Initiation of any topical drug/medication for psoriasis; Initiation of any systemic therapy for psoriasis (biologic or non-biologic).

SECONDARY OUTCOMES:
Time to Psoriasis Relapse | Baseline up to Week 96(EOS)
  Time to relapse is defined as the time interval between the last administration of Tildrakizumab and the relapse of psoriasis in days.
Absolute Psoriasis Area and Severity Index (PASI) Scores | Baseline, Weeks 12, 24, 36, 48, 60, 72, 84 and Week 96/ End of study (EOS)
  The PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and scaling on a scale range from 0 (no symptoms) to 4 (very marked), together with the percentage (%) of the area affected, rated on a scale from 0 (0%) to 6 (90-100%). PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 (no psoriasis) to 72 (the most severe disease).
Change from Baseline in Absolute Psoriasis Area and Severity Index (PASI) Scores | Baseline, Weeks 12, 24, 36, 48, 60, 72, 84 and Week 96/ End of study (EOS)
  The PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and scaling on a scale range from 0 (no symptoms) to 4 (very marked), together with the percentage (%) of the area affected, rated on a scale from 0 (0%) to 6 (90-100%). PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 (no psoriasis) to 72 (the most severe disease). Change from baseline will be calculated by subtracting post-dose value from baseline value.
Absolute Body Surface Area (BSA) Scores | Baseline, Weeks 12, 24, 36, 48, 60, 72, 84 and Week 96/ End of study (EOS)
  The BSA is a numerical score used to measure the total area of the body affected by psoriasis. The palm method will be applied: the participant's palm, including the five digits is used as a reference (representing approximately 1% of the total body surface area) and is used to repeatedly cover the lesions on the body. The investigator totals the number of palms required and then estimates the percentage (%) in each of the four body regions: head (including scalp) and neck (10%); upper extremities (20%); trunk (30%); and lower extremities (40%).
Change from Baseline in Absolute Body Surface Area (BSA) Scores | Baseline, Weeks 12, 24, 36, 48, 60, 72, 84 and Week 96/ End of study (EOS)
  The BSA is a numerical score used to measure the total area of the body affected by psoriasis. The palm method will be applied: the participant's palm, including the five digits is used as a reference (representing approximately 1% of the total body surface area) and is used to repeatedly cover the lesions on the body. The investigator totals the number of palms required and then estimates the percentage (%) in each of the four body regions: head (including scalp) and neck (10%); upper extremities (20%); trunk (30%); and lower extremities (40%). Change from baseline will be calculated by subtracting post-dose value from baseline value.
Absolute Dermatology Quality of Life Index (DLQI) Scores | Baseline, Weeks 12, 24, 36, 48, 60, 72, 84 and Week 96/ End of study (EOS)
  DLQI is a questionnaire to evaluate the impact on participant's quality of life due to psoriasis. It is composed of 10 items related to symptoms, feelings, daily activities, leisure, working or studying activities, personal relationships and opinions about dermatological treatment. Each item is scored from 0 (not affected at all) to 3 (very much affected). The DLQI score is the sum of the 10 individual question scores and ranges from 0 (no effect at all on participant's life) to 30 (extremely large effect on participant's life), with lower scores indicating better quality of life.
Absolute Dermatology Quality of Life Index Scoring Modification (DLQI-R) Scores | Baseline, Weeks 12, 24, 36, 48, 60, 72, 84 and Week 96/ End of study (EOS)
  The DLQI-R is a scoring modification for the DLQI to better evaluate not relevant responses on the DLQI that could lead to underestimation of the impact on quality of life. DLQI-R is a scoring modification involves multiplying the original DLQI score by a conversion factor that increases with the number of not relevant responses.
Change from Baseline in Absolute Dermatology Quality of Life Index (DLQI) Scores | Baseline, Weeks 12, 24, 36, 48, 60, 72, 84 and Week 96/ End of study (EOS)
  DLQI is a questionnaire to evaluate the impact on participant's quality of life due to psoriasis. It is composed of 10 items related to symptoms, feelings, daily activities, leisure, working/studying activities, personal relationships & opinions about dermatological treatment. Each item is scored from 0 (not affected at all) to 3 (very much affected). The DLQI score is the sum of the 10 individual question scores & ranges from 0 (no effect at all on participant's life) to 30 (extremely large effect on participant's life), with lower scores indicating better quality of life. Change from baseline will be calculated by subtracting post-dose value from baseline value.
Change from Baseline in Absolute Dermatology Quality of Life Index Scoring Modification (DLQI-R) Scores | Baseline, Weeks 12, 24, 36, 48, 60, 72, 84 and Week 96/ End of study (EOS)
  DLQI-R is a scoring modification for the DLQI to better evaluate not relevant responses on the DLQI that could lead to underestimation of the impact on quality of life. DLQI-R, a scoring modification involves multiplying the original DLQI score by a conversion factor that increases with the number of not relevant responses. Change from baseline will be calculated by subtracting post-dose value from baseline value.
Absolute Physician's Global Assessment (PGA) Scores | Baseline, Weeks 12, 24, 36, 48, 60, 72, 84 and Week 96/ End of study (EOS)
  The PGA is used to assess the overall severity of the psoriasis lesions at the time of evaluation. Overall lesions will be graded for erythema, induration, and scale based on 6-point scale ranging from 0 (clear) to 5 (severe). The sum of 3 scales will be divided by 3 to obtain final PGA score.
Change from Baseline in Absolute Physician Global Assessment (PGA) Scores | Baseline, Weeks 12, 24, 36, 48, 60, 72, 84 and Week 96/ End of study (EOS)
  The PGA is used to assess the overall severity of the psoriasis lesions at the time of evaluation. Overall lesions will be graded for erythema, induration, and scale based on 6-point scale ranging from 0 (clear) to 5 (severe). The sum of 3 scales will be divided by 3 to obtain final PGA score. Change from baseline will be calculated by subtracting post-dose value from baseline value.
Absolute Nail Physician Global Assessment (nPGA) Scores | Baseline, Weeks 12, 24, 36, 48, 60, 72, 84 and Week 96/ End of study (EOS)
  The nPGA is a 5-point scale ranging from 0 (clear) to 4 (severe), where higher score indicates severe nail psoriasis lesions. Only in participants with nail involvement the nPGA assessment will be performed.
Change from Baseline in Absolute Nail Physician Global Assessment (nPGA) Scores | Baseline, Weeks 12, 24, 36, 48, 60, 72, 84 and Week 96/ End of study (EOS)
  The nPGA is a 5-point scale ranging from 0 (clear) to 4 (severe), where higher score indicates severe nail psoriasis lesions. Only in participants with nail involvement the nPGA assessment will be performed. Change from baseline will be calculated by subtracting post-dose value from baseline value.
Absolute Scalp Physician Global Assessment (scPGA) Scores | Baseline, Weeks 12, 24, 36, 48, 60, 72, 84 and Week 96/ End of study (EOS)
  The scPGA score is used to assess the average severity of scalp psoriasis lesions. The scPGA is also 5-point scale ranging from 0 (clear) to 4 (severe), where higher score indicates severe scalp psoriasis lesions. Only in participants with scalp involvement, the scPGA assessment will be performed.
Change from Baseline in Absolute Scalp Physician Global Assessment (scPGA) Scores | Baseline, Weeks 12, 24, 36, 48, 60, 72, 84 and Week 96/ End of study (EOS)
  The scPGA score is used to assess the average severity of scalp psoriasis lesions. The scPGA is also 5-point scale ranging from 0 (clear) to 4 (severe), where higher score indicates severe scalp psoriasis lesions. Only in participants with scalp involvement, the scPGA assessment will be performed. Change from baseline will be calculated by subtracting post-dose value from baseline value.
Absolute Pain-Numeric Rating Scale (Pain-NRS) and Pruritus-Numeric Rating Scale (Pruritus-NRS) Scores | Baseline, Weeks 12, 24, 36, 48, 60, 72, 84 and Week 96/ End of study (EOS)
  Both Pain-NRS and Pruritus-NRS are a unidimensional segmented numeric version of the visual analog scale in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of pain or pruritus. The 11-point numeric scale of NRS ranges from 0 to 10, describing pain severity extremes scale 0 (no pain) to 10 (worst imaginable pain) and pruritus-severity extremes scale 0 (no pruritis) to 10 (worst imaginable pruritus), where higher scores indicates worse pain and pruritus.
Change from Baseline in Absolute Pain- and Pruritus-Numeric Rating Scale (NRS) Scores | Baseline, Weeks 12, 24, 36, 48, 60, 72, 84 and Week 96/ End of study (EOS)
  Both Pain-NRS and Pruritus-NRS are a unidimensional segmented numeric version of the visual analog scale in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of pain or pruritus. The 11-point numeric scale of NRS ranges from 0 to 10, describing pain severity extremes scale 0 (no pain) to 10 (worst imaginable pain) and pruritus-severity extremes scale 0 (no pruritis) to 10 (worst imaginable pruritus), where higher scores indicates worse pain and pruritus. Change from baseline will be calculated by subtracting post-dose value from baseline value.
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to Week 96/ End of study (EOS)
  An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An SAE is any untoward medical occurrence that at any dose: results in death, or is life threatening, or requires in participant hospitalization or prolongation of existing hospitalization, or results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is any other medically important event.
Number of Participants with Clinically Significant Abnormalities in Physical Examination | Baseline up to Week 96/ End of study (EOS)
  Physical Examination includes measuring height, weight, body mass index, waist circumference (cm), and waist hip ratio.
Number of Participants with Clinically Significant Change from Baseline in Vital Signs | Baseline up to Week 96/ End of study (EOS)
  Following vital signs with clinically significant observation will be measured as safety variables: diastolic and systolic blood pressure, heart rate, respiratory rate and body temperature. Change from baseline will be calculated by subtracting post-dose value from baseline value.
Number of Participants with Clinically Significant Change from Baseline in Laboratory Parameters | Baseline up to Week 96/ End of study (EOS)
  Clinically Significant hematology and biochemical parameters will be assessed. Change from baseline will be calculated by subtracting post-dose value from baseline value.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Almirall, SAS
Locations (3):
- Poland (3):
  - Site 0003, Lodz
  - Site 0001, Wroclaw
  - Site 0002, Wroclaw